CLINICAL TRIAL: NCT06745440
Title: Belgian Infective Endocarditis Registry
Acronym: BIER
Status: Not yet recruiting | Type: Observational
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Other Study IDs: 24398_BIER
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The objective of this prospective observational registry is to study patients di-agnosed with infective endocarditis (IE) and to gather comprehensive long-term outcome data, including mortality rates and IE-related complications (e.g., thromboembolic events, (hospitalization for) heart failure, valve surgery and IE recurrence) at one, three-, and five-years post-enrollment. Additionally, the registry will document epidemiological characteristics, clinical presentation at baseline, biochemical and microbiological profiles, relevant comorbidities and risk factors, diagnostic strategies, and therapeutic interventions, including an-timicrobial therapy and surgical procedures.

ELIGIBILITY:
> 18 yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Infective endocarditis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2032-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 5-years

IPD SHARING:
Plan to Share IPD: Undecided